CLINICAL TRIAL: NCT06115928
Title: Effects of VIRTUal reALity on Rehabilitation in Patients With Heart Failure: a Protocol for a Randomized Controlled Trial
Brief Title: Effects of Virtual Reality on Rehabilitation in Patients With Heart Failure
Acronym: VIRTUAL-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valentina Micheluzzi (Other)
Responsible Party: Sponsor-Investigator, Valentina Micheluzzi, MSN, RN, Azienda Ospedaliero Universitaria di Sassari
Organization: Azienda Ospedaliero Universitaria di Sassari (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOSassari
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure; Reduced Ejection Fraction
Keywords: heart failure; cardiac rehabilitation; virtual reality; treatment adherence and compliance; randomized controlled trial
MeSH Terms: conditions — Heart Failure; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): Patients will undergo cardiac rehabilitation for 30-minute each sessions, twice a week for one month with virtual reality.
  Interventions: Device: Virtual reality
- control group (No Intervention): Patients will undergo cardiac rehabilitation for 30-minute each sessions, twice a week for one month on standard care (without virtual reality)

INTERVENTIONS:
Device: Virtual reality — Participants will perform cardiac rehabilitation with hardware-type technology consisting of a PICO 4® head mounted display (HMD) headset and the software TREADMILL XR®.
  Arms: interventional group

SUMMARY:
Background. To improve symptoms and reduce poor outcomes related to heart failure (HF), international guidelines recommend cardiac rehabilitation (CR), particularly for those with a reduced ejection fraction. Unfortunately, patient adherence to rehabilitation programs remains suboptimal, with dropouts ranging from 15.4 to 63.3%. An innovative and promising intervention that could improve adherence to rehabilitation is virtual reality (VR). This study aims to evaluate the effects of VR in patients with HF undergoing CR in terms of adherence (primary outcome), functional capacity, perceived exertion, angina, quality of life, heart rate, oxygen saturation, blood pressure, maximum oxygen uptake, minute ventilation/carbon dioxide production slope, oxygen pulse, blood values of NT-proBNP and rehospitalization rates due to HF (secondary outcomes).

Methods. A randomized controlled trial will be conducted in a sample of 80 patients referred to CR. Participants will be enrolled in a cardiological rehabilitation unit of a large university hospital in Italy and randomized (1:1) to the experimental intervention consisting of CR performed with high-quality immersive VR with PICO 4® Head Mounted Display headset and TREADMILL XR® software (Arm 1) or standard CR (Arm 2). Patients will receive 30-minute CR sessions twice a week for one month.

Results. Significant improvements in primary and secondary outcomes are expected in patients in the intervention group.

Conclusions. If proven to be effective, VR could be an innovative, safe, and easy digital health intervention to improve adherence to CR in patients with HF, as well as important clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years;
* clinically stable chronic HF diagnosis with left ventricular ejection fraction (LVEF) < 40%

Exclusion Criteria:

* conditions that exclude exercise training (e.g., bone fractures);
* conditions that exclude VR use of VR (e.g., blindness and deafness
* severe cognitive impairment, documented with a score of 0 - 4 on the Six-item Screener;
* end-stage renal disease requiring dialysis;
* ascertained advanced pneumopathies;
* active neoplasms;
* rheumatic diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
adherence to cardiac rehabilitation | after 4 weeks
  adherence to cardiac rehabilitation measured as the number of sessions performed, compared to the scheduled sessions expressed as a percentage

SECONDARY OUTCOMES:
Functional capacity | at baseline, after 4 and 8 weeks
  functional capacity in meters with the six minutes walking test
Perceived exertion | at baseline, after 4 and 8 weeks
  with Borg rating of perceived exertion which captures physical activity intensity levels related to heart rate during exercise. The rate is multiplied by 10 to determine the ideal heart rate during aerobic exercise. The Borg scale score ranges from 6 to 20 corresponding to "no effort" and "maximum effort", respectively, equating a minimum of 20% to a max of 100% effort.
Angina | at baseline, after 4 and 8 weeks
  with Canadian Cardiovascular Society (CCS) grading of angina.The CCS classification system employs four grades ranging from I (no physical activity limitation) to IV (inability to perform any physical activity without discomfort).
heart rate | at baseline, after 4 and 8 weeks
  digital monitor
blood pressure | at baseline, after 4 and 8 weeks
  digital monitor
oxygen saturation | at baseline, after 4 and 8 weeks
  digital monitor
Maximal oxygen uptake | at baseline and after 8 weeks
  CPET parameters
Minute ventilation/carbon dioxide production slope | at baseline and after 8 weeks
  CPET parameters
oxygen pulse | at baseline and after 8 weeks
  CPET parameters
NT-probnp | at baseline and after 8 weeks
  blood values
HF-related rehospitalization | after 8 weeks from the stard of the study
  number of rehopedalization related to heart failure
Quality of life of patients with heart failure | at baseline, after 4 and 8 weeks
  with Kansas City Cardiomyopathy Questionnaire (KCCQ) which consists of 23 items to assess physical function, symptoms, social function, self-efficacy and quality of life of patients. KCCQ scores range from 0 to 100 and the scores represent health status as follows: from 0 to 24, very poor to poor; 25 to 49, poor to fair; 50 to 74, fair to good; and 75 to 100, good to excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Valentina Micheluzzi, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Edelmann F, Gelbrich G, Dungen HD, Frohling S, Wachter R, Stahrenberg R, Binder L, Topper A, Lashki DJ, Schwarz S, Herrmann-Lingen C, Loffler M, Hasenfuss G, Halle M, Pieske B. Exercise training improves exercise capacity and diastolic function in patients with heart failure with preserved ejection fraction: results of the Ex-DHF (Exercise training in Diastolic Heart Failure) pilot study. J Am Coll Cardiol. 2011 Oct 18;58(17):1780-91. doi: 10.1016/j.jacc.2011.06.054. PMID 21996391
- [Background] Nolte K, Herrmann-Lingen C, Wachter R, Gelbrich G, Dungen HD, Duvinage A, Hoischen N, von Oehsen K, Schwarz S, Hasenfuss G, Halle M, Pieske B, Edelmann F. Effects of exercise training on different quality of life dimensions in heart failure with preserved ejection fraction: the Ex-DHF-P trial. Eur J Prev Cardiol. 2015 May;22(5):582-93. doi: 10.1177/2047487314526071. Epub 2014 Mar 13. PMID 24627449
- [Background] Taylor RS, Long L, Mordi IR, Madsen MT, Davies EJ, Dalal H, Rees K, Singh SJ, Gluud C, Zwisler AD. Exercise-Based Rehabilitation for Heart Failure: Cochrane Systematic Review, Meta-Analysis, and Trial Sequential Analysis. JACC Heart Fail. 2019 Aug;7(8):691-705. doi: 10.1016/j.jchf.2019.04.023. Epub 2019 Jul 10. PMID 31302050
- [Background] Dunbar-Jacob J, Erlen JA, Schlenk EA, Ryan CM, Sereika SM, Doswell WM. Adherence in chronic disease. Annu Rev Nurs Res. 2000;18:48-90. PMID 10918932
- [Background] Resurreccion DM, Moreno-Peral P, Gomez-Herranz M, Rubio-Valera M, Pastor L, Caldas de Almeida JM, Motrico E. Factors associated with non-participation in and dropout from cardiac rehabilitation programmes: a systematic review of prospective cohort studies. Eur J Cardiovasc Nurs. 2019 Jan;18(1):38-47. doi: 10.1177/1474515118783157. Epub 2018 Jun 18. PMID 29909641
- [Background] Weiss PL, Kizony R, Feintuch U, Katz N. Virtual Reality in neurorehabilitation. In: Selzer M, Clarke S, Cohen L, Duncan P, Gage F, editors. Neural Repair and Rehabilitation. Cambridge; 2006. p. 182-97.
- [Background] Keshner EA, Weiss PT. Introduction to the special issue from the proceedings of the 2006 International Workshop on Virtual Reality in Rehabilitation. J Neuroeng Rehabil. 2007 Jun 6;4:18. doi: 10.1186/1743-0003-4-18. PMID 17553159
- [Background] Basso Moro S, Bisconti S, Muthalib M, Spezialetti M, Cutini S, Ferrari M, Placidi G, Quaresima V. A semi-immersive virtual reality incremental swing balance task activates prefrontal cortex: a functional near-infrared spectroscopy study. Neuroimage. 2014 Jan 15;85 Pt 1:451-60. doi: 10.1016/j.neuroimage.2013.05.031. Epub 2013 May 17. PMID 23684867
- [Background] Burrai F, Othman S, Brioni E, Micheluzzi V, Luppi M, Apuzzo L, Delli Zotti GB, La Manna G. Effects of Virtual Reality in Patients Undergoing Dialysis: Study Protocol. Holist Nurs Pract. 2019 Nov/Dec;33(6):327-337. doi: 10.1097/HNP.0000000000000330. PMID 31045610
- [Background] Meijer HA, Graafland M, Goslings JC, Schijven MP. Systematic Review on the Effects of Serious Games and Wearable Technology Used in Rehabilitation of Patients With Traumatic Bone and Soft Tissue Injuries. Arch Phys Med Rehabil. 2018 Sep;99(9):1890-1899. doi: 10.1016/j.apmr.2017.10.018. Epub 2017 Nov 11. PMID 29138050
- [Background] Pacheco TBF, de Medeiros CSP, de Oliveira VHB, Vieira ER, de Cavalcanti FAC. Effectiveness of exergames for improving mobility and balance in older adults: a systematic review and meta-analysis. Syst Rev. 2020 Jul 18;9(1):163. doi: 10.1186/s13643-020-01421-7. PMID 32682439
- [Background] Alfieri FM, da Silva Dias C, de Oliveira NC, Battistella LR. Gamification in Musculoskeletal Rehabilitation. Curr Rev Musculoskelet Med. 2022 Dec;15(6):629-636. doi: 10.1007/s12178-022-09797-w. Epub 2022 Oct 27. PMID 36301514
- [Background] Doumas I, Everard G, Dehem S, Lejeune T. Serious games for upper limb rehabilitation after stroke: a meta-analysis. J Neuroeng Rehabil. 2021 Jun 15;18(1):100. doi: 10.1186/s12984-021-00889-1. PMID 34130713
- [Background] Cikajlo I, Peterlin Potisk K. Advantages of using 3D virtual reality based training in persons with Parkinson's disease: a parallel study. J Neuroeng Rehabil. 2019 Oct 17;16(1):119. doi: 10.1186/s12984-019-0601-1. PMID 31623622
- [Background] Freeman D, Reeve S, Robinson A, Ehlers A, Clark D, Spanlang B, Slater M. Virtual reality in the assessment, understanding, and treatment of mental health disorders. Psychol Med. 2017 Oct;47(14):2393-2400. doi: 10.1017/S003329171700040X. Epub 2017 Mar 22. PMID 28325167
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768
- [Background] Xue J, Chiu HFK, Liang J, Zhu T, Jiang Y, Chen S. Validation of the Six-Item Screener to screen for cognitive impairment in primary care settings in China. Aging Ment Health. 2018 Apr;22(4):453-457. doi: 10.1080/13607863.2017.1280768. Epub 2017 Feb 1. PMID 28145741
- [Background] Uszko-Lencer NHMK, Mesquita R, Janssen E, Werter C, Brunner-La Rocca HP, Pitta F, Wouters EFM, Spruit MA. Reliability, construct validity and determinants of 6-minute walk test performance in patients with chronic heart failure. Int J Cardiol. 2017 Aug 1;240:285-290. doi: 10.1016/j.ijcard.2017.02.109. Epub 2017 Feb 28. PMID 28377186
- [Background] Day ML, McGuigan MR, Brice G, Foster C. Monitoring exercise intensity during resistance training using the session RPE scale. J Strength Cond Res. 2004 May;18(2):353-8. doi: 10.1519/R-13113.1. PMID 15142026
- [Background] Campeau L. The Canadian Cardiovascular Society grading of angina pectoris revisited 30 years later. Can J Cardiol. 2002 Apr;18(4):371-9. PMID 11992130
- [Background] Long L, Anderson L, Dewhirst AM, He J, Bridges C, Gandhi M, Taylor RS. Exercise-based cardiac rehabilitation for adults with stable angina. Cochrane Database Syst Rev. 2018 Feb 2;2(2):CD012786. doi: 10.1002/14651858.CD012786.pub2. PMID 29394453
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Burrai F, Ortu S, Marinucci M, De Marinis MG, Piredda M. Effectiveness of Immersive Virtual Reality in People with Cancer Undergoing Antiblastic Therapy: A Randomized Controlled Trial. Semin Oncol Nurs. 2023 Aug;39(4):151470. doi: 10.1016/j.soncn.2023.151470. Epub 2023 Jul 16. PMID 37455151
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Savarese G, Becher PM, Lund LH, Seferovic P, Rosano GMC, Coats AJS. Global burden of heart failure: a comprehensive and updated review of epidemiology. Cardiovasc Res. 2023 Jan 18;118(17):3272-3287. doi: 10.1093/cvr/cvac013. PMID 35150240